CLINICAL TRIAL: NCT06498102
Title: Six Weeks of Time-restricted Feeding Improves Basal Fat Oxidation and Body Composition But Not Fat Oxidation During Exercise in Young Males: A Randomized Controlled Trial
Brief Title: Time-restricted Feeding Improves Basal Fat Oxidation and Body Composition But Not Fat Oxidation During Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Muhammed Mustafa Atakan, Associate Professor of Exercise Physiology, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HU-SB-HA-02
Record Dates: First submitted 2024-06-21; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Dietary Exposure
Keywords: Diet; Intermittent Fasting; Exercise; Metabolism
MeSH Terms: conditions — Intermittent Fasting; Motor Activity

STUDY DESIGN:
Intervention Model Description: Two groups: Control (n=17) and time-restricted feeding (TRF) group (n=17)
  Thirty-four healthy recreationally active males who habitually undergo cycling, running, soccer 2-3 times per week volunteered to participate in this randomized controlled study.
Who Masked: Participant
Masking Description: Participants were randomly divided into a control (n=17) and time-restricted feeding (TRF) group (n=17).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time Restricted Feeding Group (Experimental): Thirty-one healthy, young males (age: 27.5±6 years, body mass: 76.5±8.4 kg, and maximal oxygen uptake [V̇O2max]: 43.9±6.6 mL/kg/min) were randomly assigned to either TRF (n=14) or control group (n=17). TRF group followed an 16:8 intermittent fasting diet program for 6 weeks. Body composition, insulin sensitivity, resting substrate oxidation, and fat oxidation during cycling at 40% V̇O2max were assessed before and after the diet program.
  Interventions: Other: Intermittent Fasting: Time Restricted Feeding During 6 Weeks
- Control Group (No Intervention): Control group maintained their existing dietary habits during the 6 weeks. Body composition, insulin sensitivity, resting substrate oxidation, and fat oxidation during cycling at 40% V̇O2max were assessed before and after the program.

INTERVENTIONS:
Other: Intermittent Fasting: Time Restricted Feeding During 6 Weeks — Thirty-one healthy, young males (age: 27.5±6 years, body mass: 76.5±8.4 kg, and maximal oxygen uptake [V̇O2max]: 43.9±6.6 mL/kg/min) were randomly assigned to either TRF (n=14) or control group (n=17). TRF group followed an 16:8 intermittent fasting diet program for 6 weeks. Body composition, insulin sensitivity, resting substrate oxidation, and fat oxidation during cycling at 40% V̇O2max were assessed before and after the diet program.
  Arms: Time Restricted Feeding Group

SUMMARY:
Time-restricted feeding is one of the IF models with significant advantages beyond other IF models, such as simplicity and flexibility, where individuals limit their eating window to specific hours of the day, with a fasting period of at least 12 hours. Ample evidence in humans suggests that prolonged daily cycles of feeding and fasting when aligned with the circadian rhythm, as in the TRF regimen, can alleviate metabolic diseases. Furthermore, research supports a range of health benefits associated with TRF programs in diverse populations, including improvements in body composition and insulin sensitivity, appetite regulation, and achieving a more balanced hunger sensation. Moreover, adopting a 6-hour eating window followed by an 18-hour fasting period can elicit a metabolic shift from relying on glucose to utilizing ketones for energy, which is associated with extended lifespan and a reduced risk of various diseases including type 2 diabetes and obesity. This study aimed to determine the effect of a 6-week TRF on resting and exercise substrate oxidation and changes in blood markers linked to cardiometabolic health.

DETAILED DESCRIPTION:
The aim of this study was to determine the effects of a 6-week TRF program on resting and exercise substrate oxidation, and examine changes in body composition and blood markers linked to cardiometabolic health in recreationally active young males. It was hypothesized that compared to controls, TRF would improve body composition, blood markers associated with cardiometabolic health, and increase substrate oxidation during rest and exercise.

Experimental approach to the problem:

Participants reported to the laboratory on 4 separate occasions. Initially, a familiarization session for V̇O2max testing was conducted on a cycle ergometer. In the second visit, participants repeated V̇O2max test to determine their cardiorespiratory fitness, and this test created the intensity for the submaximal exercise test. A minimum of 48 hours after the V̇O2max test and an overnight fast, body composition, resting metabolic rate (RMR), and substrate oxidation during submaximal exercise were assessed. All measurements were performed between 08:00 a.m. and 12:00 noon in order to eliminate the effect of circadian rhythm. Subsequently, participants were randomly assigned to either TRF or control group. The TRF group received comprehensive nutrition education from a dietitian and was directed to adhere to the 16:8 program for 6 weeks, limiting their eating window to 8 hours daily, while the control group was asked to maintain their eating habits. To assess participant quality of life, the 12-item Short Form Health Survey (SF-12) developed by Ware et al. was administered before and after the 6-week intervention period (38). All participants were asked to maintain their daily physical activity levels throughout the study. A 7-day food diary was completed by all participants at study initiation and during the third and sixth week. After completing the six-week program, all participants underwent post-tests identical to the pre-tests. Venous blood samples were collected from all participants following an overnight fast at baseline and after 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy recreationally active males who habitually undergo cycling, running, soccer 2-3 times per week volunteered to participate in this randomized controlled study.

Exclusion Criteria:

* Acute or chronic disease
* Taking any drug or supplements known to affect metabolism
* currently following time-restricted diets
* had lost more than 10% of their weight in the last 3 months before participated the study

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 34 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Measurement of body composition (in kg) with Dual-energy X-ray absorptiometry (DXA) | 9 months
  All participants underwent a whole-body composition scan with light clothing to measure total body mass (kg), fat mass (kg), fat-free mass (kg), and lean body mass (kg), with an automatically chosen scanning mode by the DXA machine (Lunar Prodigy Pro Narrow Fan Beam (4.5º), GE Health Care, Madison, Wisconsin, USA).
V̇O2max measurement | 9 months
  Participants' V̇O2max was determined using an incremental exercise test on a cycle ergometer (COSMED E 200, Rome, Italy). The test consisted of 2 minutes of cycling at 60 W, 120 W, and 150 W, respectively. Afterward, the workload increased by 30 W every minute until voluntary exhaustion. Heart rate (HR) was continuously recorded during the test using a HR monitor. Breath-by-breath expired air was acquired throughout the test using an online gas analysis system (Quark Cardio Pulmonary Exercise Testing, COSMED, Rome, Italy). The gas analyzer was periodically calibrated according to the manufacturer's procedures prior to each test. The recorded value for V̇O2max was the highest achieved over a 30-second sampling period.
Measurement of resting metabolic rate (RMR) | 9 months
  RMR was determined using a breath-by-breath indirect system (CPET, Rome, Italy). Participants were required to fast for 10-12 hours before testing and limit physical activity on their way to the laboratory. Upon arriving at the laboratory, participants rested in a dimly lit, temperature-controlled room in a supine position, and were instructed to relax without falling asleep. The protocol involved a 20-minute rest in the supine position, followed by a 15-minute period of respiratory gas analysis. During the respiratory gas analysis, oxygen uptake and carbon dioxide output were measured using a breath-by-breath system with a breathing mask connected to a pre-calibrated computerized gas analyzer.
Calculation of resting substrate oxidation | 9 months
  We used the respiratory data (oxygen and carbon dioxide) collected during the RMR measurement to calculate resting fat (g/min) and resting carbohydrate oxidation (g/min) using the Frayn equation, as follows:
  Fat oxidation (g/min) = 1,67 × V̇O2 (L/min) - 1,67 × V̇CO2 (L/min) CHO oxidation (g/min) = 4,55 × V̇CO2 (L/min) - 3,21 × V̇O2 (L/min)
Measurement of substrate oxidation during submaximal exercise | 9 months
  A few minutes after RMR assessment, participants cycled for 30 minutes at a workload corresponding to 40% of their pre-determined V̇O2max on cycle ergometer (COSMED E 200, Italy) before and after the TRF program. The test commenced with a 3-minute warm-up at 60 W. V̇O2 and V̇CO2 during the test were recorded using an online gas analysis system (Quark Cardio Pulmonary Exercise Testing, COSMED, Rome, Italy). Fat oxidation and CHO oxidation were computed utilizing the equation proposed by Jeukendrup and Wallis.
Food Diary | 9 months
  All participants completed a 7-day food diary at the commencement of the study, during the third week, and at the end of the sixth week to assess any potential changes in participant dietary habits. An experienced dietician determined the portion size with household units, such as cups, pieces, or plates. In addition, the ingredients of mixed dishes were specified, and product name and standard weights of food items were used to calculate serving sizes. All the results were calculated and analyzed by the same experienced dietician using Nutrition Information System (BEBIS 6.1, Dr. J. Erhardt, Stutgart, Hohenheim, Germany).
Time Restricted Feeding | 9 months
  The TRF group received detailed nutrition education before the TRF program, and was instructed to follow the 16:8 program for six weeks, limiting their eating window to 8 hours daily (10:00 to 18:00 or alternatively 11:00 to 19:00), during which no calorie restriction was applied. During the 16-hour fasting window, the TRF group was asked to avoid calorie-containing foods and beverages. All participants in both groups were contacted twice a week to monitor dietary compliance in the TRF group and to maintain their existing eating habits in the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Atakan, PhD, Study Director — Hacettepe University; Hale Aktaş, MSc, Study Chair — Hacettepe University; Hüseyin Turnagöl, Professor, Principal Investigator — Hacettepe University; Nazan Koşar, Proffesor, Study Chair — Hacettepe University; Zeynep Ergün, BsC, Study Chair — Hacettepe University
Locations (1):
- Faculty of Sports Science, Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stratton MT, Tinsley GM, Alesi MG, Hester GM, Olmos AA, Serafini PR, Modjeski AS, Mangine GT, King K, Savage SN, Webb AT, VanDusseldorp TA. Four Weeks of Time-Restricted Feeding Combined with Resistance Training Does Not Differentially Influence Measures of Body Composition, Muscle Performance, Resting Energy Expenditure, and Blood Biomarkers. Nutrients. 2020 Apr 17;12(4):1126. doi: 10.3390/nu12041126. PMID 32316561
- [Background] Mattson MP, Allison DB, Fontana L, Harvie M, Longo VD, Malaisse WJ, Mosley M, Notterpek L, Ravussin E, Scheer FA, Seyfried TN, Varady KA, Panda S. Meal frequency and timing in health and disease. Proc Natl Acad Sci U S A. 2014 Nov 25;111(47):16647-53. doi: 10.1073/pnas.1413965111. Epub 2014 Nov 17. PMID 25404320
- [Background] Panda S. Circadian physiology of metabolism. Science. 2016 Nov 25;354(6315):1008-1015. doi: 10.1126/science.aah4967. PMID 27885007
- [Background] Di Francesco A, Di Germanio C, Bernier M, de Cabo R. A time to fast. Science. 2018 Nov 16;362(6416):770-775. doi: 10.1126/science.aau2095. PMID 30442801
- [Background] Atakan MM, Guzel Y, Bulut S, Kosar SN, McConell GK, Turnagol HH. Six high-intensity interval training sessions over 5 days increases maximal oxygen uptake, endurance capacity, and sub-maximal exercise fat oxidation as much as 6 high-intensity interval training sessions over 2 weeks. J Sport Health Sci. 2021 Jul;10(4):478-487. doi: 10.1016/j.jshs.2020.06.008. Epub 2020 Jun 18. PMID 32565243
- [Background] Atakan MM, Guzel Y, Shrestha N, Kosar SN, Grgic J, Astorino TA, Turnagol HH, Pedisic Z. Effects of high-intensity interval training (HIIT) and sprint interval training (SIT) on fat oxidation during exercise: a systematic review and meta-analysis. Br J Sports Med. 2022 Jul 20:bjsports-2021-105181. doi: 10.1136/bjsports-2021-105181. Online ahead of print. PMID 35859145
- [Background] Atakan MM, Kosar SN, Turnagol HH. Six Sessions of Low-volume High-intensity Interval Exercise Improves Resting Fat Oxidation. Int J Sports Med. 2022 Dec;43(14):1206-1213. doi: 10.1055/a-1905-7985. Epub 2022 Jul 20. PMID 35858638
- [Background] Xie Z, Sun Y, Ye Y, Hu D, Zhang H, He Z, Zhao H, Yang H, Mao Y. Randomized controlled trial for time-restricted eating in healthy volunteers without obesity. Nat Commun. 2022 Feb 22;13(1):1003. doi: 10.1038/s41467-022-28662-5. PMID 35194047
- [Derived] Aktas H, Atakan MM, Aktitiz S, Ergun Z, Kosar SN, Astorino TA, Turnagol HH. Six weeks of time-restricted eating improves basal fat oxidation and body composition but not fat oxidation during exercise in young males. Clin Nutr. 2025 Jul;50:92-103. doi: 10.1016/j.clnu.2025.04.022. Epub 2025 Apr 30. PMID 40382896